CLINICAL TRIAL: NCT00135161
Title: Feasibility Study of Incorporating 18F-FDG-PET Imaging in Radiotherapy for Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Belgian Federation Against Cancer (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003/202
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Head and Neck Neoplasms
Keywords: neoplasms (squamous cell carcinoma of the head and neck region)
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intensity modulated radiation therapy (IMRT). (Experimental)
  Interventions: Procedure: FDG-PET-based dose escalation using intensity modulated radiation therapy (IMRT).

INTERVENTIONS:
Procedure: FDG-PET-based dose escalation using intensity modulated radiation therapy (IMRT). — FDG-PET-based dose escalation using intensity modulated radiation therapy (IMRT).

SUMMARY:
The purpose of this trial is to study fluorodeoxyglucose-positron emission tomography (FDG-PET)-based dose escalation using intensity modulated radiation therapy (IMRT).

DETAILED DESCRIPTION:
The dose escalation, based on the FDG-PET signal, is incorporated in the first ten fractions of the radiotherapeutic treatment. The total amount of fractions is 32, equal to a standard radiotherapeutic treatment for these types of cancers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a proven histological squamous cell carcinoma of the larynx (only T3-4 NO or Tany N+), hypopharynx, oropharynx
* Patients who did not undergo surgery for the primary tumor location
* Patients with a Karnofsky performance score of 70% or more
* Written informed consent for participation in this trial

Exclusion Criteria:

* Other malignancy except for non-melanoma skin cancer
* Prior irradiation to the head and neck region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2003-09 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Acute toxicity during radiotherapy until 3 months after the end of the radiotherapy | until 3 months after the end of the radiotherapy
Observation of chronic toxicity | until 3 months after the end of the radiotherapy

SECONDARY OUTCOMES:
Therapy response (2-4 months after end of radiotherapy) | 2-4 months after end of radiotherapy
Local control at 2 years | at 2 years
Pattern of recurrence | at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Neve, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be